CLINICAL TRIAL: NCT05276687
Title: Efficacy of Diluted Betadine vs Antibiotic Installation Before Surgical Wound Closure in Prevention of Post Cardiac Surgery Wound Infection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman Hamed Ahmed, Resident doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: diluted betadine vs antibiotic
Record Dates: First submitted 2022-03-03; First posted 2022-03-11 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Surgical Wound Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Povidone-Iodine; Vancomycin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Diluted betadine (Experimental)
  Interventions: Drug: Betadine
- Powdered vancomycin (Experimental)
  Interventions: Drug: Vancomycin
- No intervention (No Intervention)

INTERVENTIONS:
Drug: Betadine — Wound irrigation
  Arms: Diluted betadine
Drug: Vancomycin — instillation in the wound
  Arms: Powdered vancomycin

SUMMARY:
1. Infection control and health-care-associated infections and Safety of medical service providers
2. Evidence based management of common medical and surgical problems

DETAILED DESCRIPTION:
Surgical wound infection is the presence of replicating micro-organisms within a wound of a surgery leading to host injury. Superficial sternal wound infection (SSWI) is the infection that affects the skin and subcutaneous tissues and the pectoralis fascia(1,2). Deep sternal wound infection (DSWI) is the infection affecting muscle layer and the bony sternum, it is one of the most complex and potentially devastating complications following median sternotomy in cardiac surgery with a significant impact on both patient prognosis and hospital budgets, despite of many advances in prevention, it is still remaining significant, and ranges between 0.5% and 6.8%(2), with in-hospital mortality between 7% and 35%. moreover, mid- and long- term survival is significantly reduced in patients that have experienced DSWI(3). Sternal dehiscence is the process of separation of bony sternum which is often accompanied by mediastinits(4). Although prevention of infection following arthroplasty requires a multifaceted approach, the use of intraoperative irrigation is an important component of any protocol. Recent clinical practice guidelines from the Centers for Disease Control, World Health Organization, and International Consensus Meeting on Musculoskeletal Infection advocate the use of a dilute povidone-iodine solution prior to wound closure. This experience suggests that this practice is safe, inexpensive, and easily implemented(5). The present study is going to discuss the effect of dilute povidone-iodine irrigation vs vancomycine irrigation intraoperative in prevention of postoperative infection after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* age from 1 to 65 years, primary or redo cases

Exclusion Criteria:

* diabetic patients

Ages: 1 Year to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Superficial wound infection | Within 20 days
Deep wound infection | Within 20 days

SECONDARY OUTCOMES:
Healing of sternum ( within 2 months) | 20 days to 60 days

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cotogni P, Barbero C, Rinaldi M. Deep sternal wound infection after cardiac surgery: Evidences and controversies. World J Crit Care Med. 2015 Nov 4;4(4):265-73. doi: 10.5492/wjccm.v4.i4.265. eCollection 2015 Nov 4. PMID 26557476
- [Background] Singh K, Anderson E, Harper JG. Overview and management of sternal wound infection. Semin Plast Surg. 2011 Feb;25(1):25-33. doi: 10.1055/s-0031-1275168. PMID 22294940
- [Background] Kotnis-Gaska A, Mazur P, Olechowska-Jarzab A, Stanisz A, Bulanda M, Undas A. Sternal wound infections following cardiac surgery and their management: a single-centre study from the years 2016-2017. Kardiochir Torakochirurgia Pol. 2018 Jun;15(2):79-85. doi: 10.5114/kitp.2018.76472. Epub 2018 Jun 25. PMID 30069187
- [Background] Asghar A, Talha KM, Amanullah M, Shahabuddin S. Comparison of figure of eight and traditional simple wire closure method to prevent dehiscence after sternal closure. J Pak Med Assoc. 2020 Nov;70(11):2001-2006. doi: 10.5455/JPMA.20135. PMID 33341848
- [Background] Goswami K, Austin MS. Intraoperative povidone-iodine irrigation for infection prevention. Arthroplast Today. 2019 May 22;5(3):306-308. doi: 10.1016/j.artd.2019.04.004. eCollection 2019 Sep. PMID 31516971